CLINICAL TRIAL: NCT07007741
Title: A Randomised Controlled Trial Study of the Effect of Fatty Liver Data Analysis and Management Software on the Effectiveness of Intervention in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Digital Therapy for Fatty Liver Disease
Acronym: DTFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-25-001
Record Dates: First submitted 2025-03-06; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-01

CONDITIONS: Steatohepatitis, Nonalcoholic; Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Software Group (Experimental): Download the Fatty Liver Data Analysis and Intervention Software and associate it with the researcher. Baseline data was collected, a health record was created, and the Weight and Lipo Meter that came with the software was linked to the software for data collection. The researcher assesses the participant through the software (on the part of the physician) and develops a diet and exercise plan based on the participant's individual circumstances. At weeks 12 and 24 after enrolment, study participants were notified of follow-up examinations to collect data on body weight, waist and hip circumference, blood tests, liver function, kidney function, blood lipids, fasting blood glucose, fasting insulin, glycated haemoglobin, abdominal ultrasound, liver transient elasticity, and body composition measurements.
  Interventions: Other: Software Group
- Life Group (No Intervention): Under the guidance of the programme specialist, the enrolled study participants collected baseline data and established health records. Professional clinicians will provide offline health education and lifestyle guidance according to the latest Chinese NAFLD prevention and treatment guidelines. At weeks 12 and 24 after enrolment, study participants were notified of follow-up examinations to collect data on body weight, waist and hip circumference, blood tests, liver function, kidney function, blood lipids, fasting blood glucose, fasting insulin, glycated haemoglobin, abdominal ultrasound, liver transient elasticity, and body composition measurements.

INTERVENTIONS:
Other: Software Group — Download the "Fatty Liver Data Analysis and Management Software", register and update your profile, connect to a scale, and associate with a researcher and dietitian. Upload meal charts and weight and body fat data every day, adjust recipes according to the patient's exercise and diet every week, and customise one-on-one Q&A according to the patient's uploaded photos every day. After enrolment, w12 and w24 were required to follow-up to complete relevant examinations and scales and collect data.
  Arms: Software Group

SUMMARY:
This study is a randomised controlled trial of the clinical application of the Fatty Liver Data Analysis and Intervention System (FLDAS) to compare the effectiveness of traditional lifestyle interventions in patients with fatty liver with digital therapies combining software and hardware devices; to validate the effectiveness of digital therapies in patients with fatty liver; and to evaluate the effectiveness of remote lifestyle (diet and exercise) interventions.

Researchers conducted a randomised controlled trial to compare the effectiveness of a traditional lifestyle intervention for patients with fatty liver with a remote lifestyle (diet and exercise) intervention combining digital therapy software and hardware devices. When the effectiveness of this programme is validated, it could help clinicians improve the efficiency of lifestyle interventions for patients with fatty liver and address the growing need for primary care for patients with fatty liver as an innovative approach to disease intervention.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD patient (CAP value >248 (dB/m))
* Age 18-65 years old, 24kg/m2 ≤ BMI ≤ 35kg/m2
* Must be able to use smartphone

Exclusion Criteria:

* Inherited metabolic or autoimmune liver disease
* Drug/toxic/alcoholic/biliary liver injury, cirrhosis or any end-stage liver disease
* Hepatic or extrahepatic malignant tumours
* Pregnant and lactating women
* Patients considered ineligible by the investigator's clinical judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduced body weight rate | Week 12 & Week 24
  The Fatty Liver Data Analysis and Intervention Software (FLADIS) was used to assist clinicians with remote data monitoring and follow-up of NAFLD patients, as well as lifestyle intervention guidance and follow-up management, and to evaluate the effectiveness of the FLADIS intervention on the degree of weight loss in patients with NAFLD.

SECONDARY OUTCOMES:
Decreased CAP Value (Indicating Reduced Liver Fat) | Week 12 & Week 24
  The Fatty Liver Data Analysis and Intervention Software (FLADlS) was used to assist clinicians with remote data monitoring and follow-up of NAFLD patients,as well as lifestye intervention guidance and follow-up management, and to evaluate the effectiveness of the FLADIS intervention in restoring NAFLD patients' Controlled Attenuation Parameter (CAP) values to normal ranges (CAP < 248 dB/m)

CONTACTS AND LOCATIONS:
Locations (1):
- XinHua Hospital Affiliated To Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No